CLINICAL TRIAL: NCT06468462
Title: WHO-recommended Periodic Presumptive Treatment Versus Doxycycline Post-Exposure Prophylaxis for STI Control Among Cisgender Men Who Have Sex With Men in Kenya
Brief Title: Periodic Presumptive Treatment vs. doxyPEP for STI Control in Kenyan MSM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Aurum Institute (Other); Nyanza Reproductive Health Society (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Partners for Health & Development in Africa (Unknown)
Responsible Party: Principal Investigator, Susan Graham, Professor: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00018588; 1R01AI179838-01 (NIH)
Record Dates: First submitted 2024-06-01; First posted 2024-06-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Gonorrhea Male; Chlamydia (Male); Syphilis Male
Keywords: gonorrhea; chlamydia; syphilis
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea; Syphilis

STUDY DESIGN:
Intervention Model Description: The proposed study is an open-label randomized controlled trial with a hybrid type 1 implementation-effectiveness component comparing each intervention (i.e., STI PPT, doxyPEP) to a common control in a 2:2:1 ratio.
  Approach for objective 1: We will conduct an open-label randomized clinical trial with 2900 participants to evaluate these two interventions versus the standard of care assigned in a 2:2:1 ratio, with 18 months of follow-up and rigorous culture-based and molecular analysis of AMR in NG at three MSM-friendly research clinics in Kenya.
  Approach for objective 2: We will use multidisciplinary science to measure the acceptability, feasibility, and safety of these two interventions, using a conceptual model based on Proctor's Implementation Science Framework.
  Approach for objective 3: Aim 1 and 2 results will inform parameters to update a stochastic model of STI transmission and cost-effectiveness analysis to project the impact of scaled-up STI PPT and doxyPEP in Kenya.
Who Masked: Outcomes Assessor
Masking Description: Aptima Combo 2 testing for NG and CT will be conducted in Mombasa on a Hologic Panther platform by experienced laboratory staff blinded to randomization assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- WHO-recommended periodic presumptive treatment (Active Comparator): Participants assigned to the STI PPT arm will be evaluated at baseline and every 3 months thereafter for STI PPT eligibility based on having had condomless anal sex and either multiple sex partners or a sex partner with an STI in the past 6 months. If eligible, they will be offered 400 mg po cefixime plus 1 gram azithromycin po under direct observation, using the same regimen as for syndromic treatment per the latest WHO recommendations.
  Interventions: Drug: WHO-recommended periodic presumptive treatment
- Doxycycline post-exposure prophylaxis (Active Comparator): Participants assigned to the doxyPEP arm will be provided with a 30-day supply of doxycycline hyclate at each quarterly visit, with refills as needed. They will have 1:1 counselling on the self-administration of 200 mg po doxycycline within 24-72 hours after condomless anal or vaginal sex as frequently as daily if indicated but not more than once daily, in accordance with the doxyPEP trial in the United States.
  Interventions: Drug: Doxycycline post-exposure prophylaxis
- Standard care (No Intervention): Participants assigned to the standard care arm will receive screening for STI symptoms at every scheduled visit and syndromic treatment with cefixime 400 mg po stat plus azithromycin 1 gram po stat under direct observation, in accordance with current Kenyan recommendations for genital and anorectal infections. This regimen will be updated if Kenyan recommendations change.

INTERVENTIONS:
Drug: WHO-recommended periodic presumptive treatment — 400 mg po cefixime plus 1 gram azithromycin po under direct observation
  Other Names: WHO PPT
  Arms: WHO-recommended periodic presumptive treatment
Drug: Doxycycline post-exposure prophylaxis — 200 mg po doxycycline within 24-72 hours after condomless anal or vaginal sex as frequently as daily
  Other Names: doxyPEP
  Arms: Doxycycline post-exposure prophylaxis

SUMMARY:
Men who have sex with men (MSM) are at high risk for gonorrhea and chlamydia in Kenya, where nucleic acid amplification testing is not feasible and most infections therefore go undiagnosed. We propose an open-label randomized clinical trial with 2900 participants assigned to WHO-recommended periodic presumptive treatment (PPT) or doxycycline post-exposure prophylaxis (doxyPEP), compared to standard syndromic treatment, with 18 months of follow-up and rigorous culture-based and molecular analysis of antimicrobial resistance in Neisseria gonorrhoeae. This work will provide critical data needed to inform guidelines and improve STI control among MSM in sub-Saharan Africa and other resource-limited settings, including modelled estimates of the health and economic impact of scaling up these two interventions on STI control among MSM and their partners in Kenya.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) are at high risk for gonorrhoea and chlamydia in Kenya, where nucleic acid amplification testing (NAAT) is not feasible, and most infections therefore go undiagnosed. In 2011, the WHO recommended periodic presumptive treatment (PPT) of Neisseria gonorrhoeae (NG) and Chlamydia trachomatis (CT) infections for MSM at high risk for HIV acquisition due to condomless anal intercourse with multiple sex partners or a recent STI exposure. More recently, trials in well-resourced settings have demonstrated the efficacy of doxycycline post-exposure prophylaxis (doxyPEP) for reducing NG, CT, and syphilis infections among high-risk MSM. The goal of this study is to evaluate the impact and cost-effectiveness of WHO-recommended PPT versus doxyPEP compared to standard syndromic treatment among Kenyan MSM. This study aims to (1) evaluate the effectiveness and impact on antimicrobial resistance in NG of WHO-recommended PPT given every 3 months and of doxy-PEP taken 24-72 hours after condomless sex for reducing STI burden among Kenyan MSM; (2) assess the acceptability, feasibility, and safety of implementing WHO-recommended PPT and doxy-PEP compared to standard care among providers and patients; and (3) model the health and economic impact of scaling up WHO-recommended STI PPT and doxyPEP compared to standard of care on STI control among MSM and their partners in Kenya. We will conduct an open-label randomized trial with 2900 participants to evaluate these two interventions versus standard care assigned in a 2:2:1 ratio, with 18 months of follow-up at three MSM-friendly research clinics in Kenya. Results will inform parameters to update a stochastic model of STI transmission and cost-effectiveness analysis to project the impact of scaled-up STI PPT and doxyPEP in Kenya. This work will provide the critical data needed to inform guidelines and improve STI control among this key population in sub-Saharan Africa and other resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* 18-29 years old
* Assigned male sex at birth
* Identifies as male (cis-gender)
* Reports condomless anal intercourse with a man in the past 6 months
* Reports multiple male sex partners OR a male sex partner with a syndromic (urethritis, proctitis, or genital ulcer disease) or laboratory-diagnosed sexually transmitted infection in the past 6 months
* Willing and able to provide written informed consent and participate in all study procedures
* Planning to remain in the study area for 18 months

Exclusion Criteria:

* Unable to understand the study purpose and procedures
* Allergy to cephalosporin (cefixime), macrolide (erythromycin or azithromycin), or tetracycline (doxycycline) class antibiotics
* Recent use of prolonged antibiotics (≥14-day course in the month before enrolment)
* Use of medications that impact cefixime, azithromycin, or doxycycline metabolism (check versus list in screening SOP)

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — identifies as male (cis-gender)
Enrollment: 2900 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with NG, CT, or early syphilis infection (combined STI outcome) | Over 18 months of follow-up at quarterly visits from the date of randomization
  The number of participants with the combined STI outcome will be determined at each visit. The combined STI outcome will be positive when any Aptima test on a pooled specimen (throat, rectal, and urine) is positive for CT or NG or any participant tests positive for early syphilis infection, defined as a positive rapid plasma reagin [RPR] in a previously negative participant or a fourfold increase in non-treponemal titres for participants with a history of syphilis.

SECONDARY OUTCOMES:
Number of participants with Neisseria gonorrhea infection | Over 18 months of follow-up at quarterly visits from the date of randomization
  The number of participants with an Aptima test on a pooled specimen (throat, rectal, and urine) positive for NG will be determined at each visit.
Number of participants with Chlamydia trachomatis infection | Over 18 months of follow-up at quarterly visits from the date of randomization
  The number of participants with an Aptima test on a pooled specimen (throat, rectal, and urine) positive for CT will be determined at each visit.
Number of participants with early syphilis infection | Over 18 months of follow-up at quarterly visits from the date of randomization
  The number of participants with early syphilis infection, defined as a positive rapid plasma reagin [RPR] in a previously negative participant or a fourfold increase in non-treponemal titres for participants with a history of syphilis, will be determined at each visit

OTHER OUTCOMES:
Number of gonorrhea infections with antimicrobial resistance mutations | Over 18 months of follow-up at quarterly visits from the date of randomization
  The number of gonorrhea infections with genetic determinants conferring resistance to cefixime, azithromycin or tetracycline resistance will be determined a each visit
Acceptability of Intervention Measure | Measured every 6 months over 18 months of follow-up from the date of randomization
  The Acceptability of Intervention Measure (4 questions rated from 0 to 4) will be assessed at baseline and every 6 months thereafter in all study arms. The "intervention" assessed will be the study arm to which the participant is assigned (i.e., presumptive treatment, doxyPEP, or standard care).
Feasibility of Intervention Measure | Measured every 6 months over 18 months of follow-up from the date of randomization
  The Feasibility of Intervention Measure (4 questions rated from 0 to 4) will be assessed at baseline and every 6 months thereafter in all study arms. The "intervention" assessed will be the study arm to which the participant is assigned (i.e., presumptive treatment, doxyPEP, or standard care).
Adverse events | Over 18 months of follow-up at quarterly visits from the date of randomization
  Number of adverse events, including social harms, reported by participants or study staff at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Graham, MD, PhD, MPH, Principal Investigator — University of Washington
Locations (3):
- Kenya (3):
  - Anza Mapema Clinic, Kisumu
  - University of Washington/Pwani Research Centre at the Ganjoni Municipal Clinic, Mombasa, Mombasa
  - TRANSFORM Clinic, Nairobi

IPD SHARING:
Plan to Share IPD: Yes
All data produced in the course of the project will be preserved and shared. The final dataset will include self-reported demographic and behavioral data from interviews with participants, clinical data from participant symptoms and focused physical exams, and laboratory data from blood and genitourinary specimens provided.
  We will share de-identified individual-participant level data. Appropriate measures such as expert determination to identify for removal any specific variables that could potentially lead to identification of individuals. Plans for data de-identification and sharing will be reflected in the informed consent forms.
  To facilitate interpretation of the data, a data dictionary describing all variables in the dataset, the study protocol, and all data collection instruments will be created, shared, and associated with the relevant datasets. Documentation and support materials will be compatible with the clinicaltrials.gov Protocol Registration Data Elements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available indefinitely from year 5 of the 5-year funded grant cycle.
Access Criteria: Due to ethical considerations, access, distribution, and reuse of the resulting scientific data will be limited to collaborations in which a formal data sharing agreement is developed and approved by the University of Washington and Kenyatta National Hospital Ethical Review Boards.

REFERENCES:
- [Derived] Graham SM, Otieno FO, Kimani J, Barrientos A, Soge OO, Sharma M, Hamilton DT, Celum C, McClelland RS, Sanders EJ. World Health Organization-Recommended Periodic Presumptive Treatment Versus Doxycycline Post-Exposure Prophylaxis for Sexually Transmitted Infection Control Among Men Who Have Sex With Men in Kenya: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2026 Jan 6;15:e81113. doi: 10.2196/81113. PMID 41494183

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT06468462/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT06468462/ICF_001.pdf